CLINICAL TRIAL: NCT07123168
Title: Effect of a Nurse-Led, Triangle-Based Hierarchical Management Model on Quality of Life, Disease-Related Knowledge, Self-Management, and Treatment Adherence in Patients Undergoing Maintenance Hemodialysis: A Randomized Controlled Trial
Brief Title: Hierarchical Management for Maintenance Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yanyan Deng (Other)
Responsible Party: Sponsor-Investigator, Yanyan Deng, Principal investigator, Shiyan Xiyuan Hospital
Organization: Shiyan Xiyuan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: surmyy2023-039
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: End-stage Renal Disease (ESRD)
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Observation Group (Triangle Hierarchical Management) (Experimental): Participants received care based on a nurse-led, Triangle Hierarchical Management model for 24 weeks. Upon enrollment, patients were stratified into high-, medium-, or low-risk tiers based on clinical, functional, and psychological criteria. Management strategies, including nurse-to-patient ratios, health education intensity, and psychological support, were tailored to the risk tier. Patients were re-evaluated weekly, and their risk classification and management plan were adjusted accordingly.
  Interventions: Behavioral: Triangle Hierarchical Management
- Active Comparator: Control Group (Routine Care) (Active Comparator): Participants received routine nursing care for 24 weeks. This included standard monitoring of laboratory parameters and vital signs, vascular access assessment, and one general health education session per month for patients and/or their families.
  Interventions: Behavioral: routine care

INTERVENTIONS:
Behavioral: Triangle Hierarchical Management — A nurse-led, risk-stratified management model where patients are categorized into high-, medium-, or low-risk tiers. High-risk patients receive intensive professional care (90%) and minimal self-management education (10%); medium-risk patients receive a balanced approach (50% each); and low-risk patients focus on self-management education (90%) with minimal professional care (10%). The intervention is delivered by trained nurses over 24 weeks.
  Arms: Experimental: Observation Group (Triangle Hierarchical Management)
Behavioral: routine care — Standard nursing management for hemodialysis patients, including monthly monitoring, routine assessments, and general health education sessions. This care does not involve risk stratification or tailored interventions.
  Arms: Active Comparator: Control Group (Routine Care)

SUMMARY:
This prospective, randomized controlled trial investigates the effectiveness of a nurse-led, Triangle Hierarchical Management model compared to routine care for patients on maintenance hemodialysis. The study aims to determine if this risk-stratified management approach improves patients' quality of life, disease-related knowledge, self-management capabilities, and treatment adherence over a 24-week period.

DETAILED DESCRIPTION:
Patients undergoing maintenance hemodialysis (MHD) face significant disease burdens, leading to poor quality of life and suboptimal self-management. Conventional nursing care often lacks individualized strategies. The "Triangle" model of chronic care management, which stratifies patients into high-, medium-, and low-risk tiers, allows for targeted allocation of healthcare resources and education. This study adapted this model for an MHD population through a Delphi consultation with experts. Eighty patients were randomized to either receive the Triangle Hierarchical Management intervention or routine care for 24 weeks. The intervention group received tailored nursing support based on their risk level, which was re-assessed weekly. The study's objective is to provide evidence on whether this structured, risk-based nursing model is superior to standard care in improving key patient-reported outcomes for the MHD population in China.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosed with uremia and receiving maintenance hemodialysis for ≥ 6 months.
* Willing to participate and provide written informed consent.

Exclusion Criteria:

* Presence of severe psychiatric, intellectual, or cognitive impairments.
* Diagnosis of severe cardiac, pulmonary, hepatic, or hematologic diseases or malignant tumors.
* Presence of a severe active infection.
* Concurrent participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life (QoL) | Baseline, 24 Weeks
  Measured using the Mandarin Chinese version of the Kidney Disease Quality of Life-Short Form (KDQOL-SF™ 1.3). The instrument assesses both kidney disease-targeted areas (KDTA) and generic health (SF-36). Scores for each domain are transformed to a 0-100 scale, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Change in Disease-Related Knowledge | Baseline, 24 Weeks
  Measured using the 24-item Hemodialysis Knowledge Questionnaire. The total score ranges from 0 to 24, with higher scores indicating greater knowledge.
Change in Self-Management Ability | Baseline, 24 Weeks
  Measured using the 20-item Hemodialysis Self-Management Instrument (HD-SMI). The total score ranges from 20 to 80, with higher scores reflecting better self-management ability.
Change in Treatment Adherence | Baseline, 24 Weeks
  Measured using the 23-item Treatment Adherence Scale for Hemodialysis Patients. The total score ranges from 23 to 115, with higher scores indicating better adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital, Hubei University of Medicine, Shiyan, Hubei, China